CLINICAL TRIAL: NCT01759199
Title: The Six-minute Stepper Test : Marker of Exercise Tolerance's Evolution During Pulmonary Rehabilitation in Patients With COPD ?
Brief Title: The Six-minute Stepper Test as an Outcome Measure of Exercise Tolerance During Pulmonary Rehabilitation in With Chronic Obstructive Pulmonary Disease (COPD) Patients(STEPPER)?
Acronym: STEPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RB 11-157 STEPPER
Record Dates: First submitted 2012-12-04; First posted 2013-01-03 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2013-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; ST6: The six minute Stepper Test; Conventional respiratory rehabilitation; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The six minute Stepper Test (Experimental): Experimental : The six minute Stepper Test with a Conventional respiratory rehabilitation
  Interventions: Procedure: Pulmonary rehabilitation assessed with six-minute walk test and six-minute stepper test

INTERVENTIONS:
Procedure: Pulmonary rehabilitation assessed with six-minute walk test and six-minute stepper test

SUMMARY:
The aim of this study is to show if the six-minute stepper test (ST6) is a sensible marker of exercise tolerance evolution during a pulmonary rehabilitation program in people with all stages of severity of Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Currently, the reference test in assessing functional capacity in COPD patients during pulmonary rehabilitation is the six-Minute Walking Test (6MWT). However, the realization of the 6MWT requires a 30m-long corridor, according to the American Thoracic Society Guidelines. Lack of sufficient space can prevent the realization of 6MWT, especially for private practitioner pulmonologists, and also in hospitals. The six-minute stepper test (ST6) which can be performed in a normal room, should be an interesting alternative.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COPD wtih all stages of severity
* Hospitalized in the pulmonary rehabilitation unit in the hospital of Morlaix, with a 3 weeks pulmonary rehabilitation course

Exclusion Criteria:

* Pneumonectomy, Lobectomy less than 6 months
* orthopedic problem
* Balance disorder
* Weight > 110kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The number of steps to The Six-minute Stepper Test (ST6) | 21 days
  Assess the difference in the number of steps in ST6 before and after pulmonary rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: FRANCIS COUTURAUD, MD,PHD, Principal Investigator — Brest University Hospital Brest,, Brittany, France 29200; CATHERINE LE BER-MOY, DR., Principal Investigator — Hospital of Morlaix Morlaix, Brittany, France 29600; CHANTAL LOCHON, DR., Principal Investigator — Hospital of Morlaix Morlaix, Brittany, France 29600
Locations (3):
- France (3):
  - Brest University Hospital, Brest, Brittany Region
  - Hospital of Morlaix, Morlaix, Brittany Region
  - Hospital of Morlaix, Morlaix, Brittany

REFERENCES:
- [Result] Pichon R, Couturaud F, Mialon P, Le Ber-Moy C, Peran L, Lochon C, Nowak E, Beaumont M. Responsiveness and Minimally Important Difference of the 6-Minute Stepper Test in Patients with Chronic Obstructive Pulmonary Disease. Respiration. 2016;91(5):367-73. doi: 10.1159/000446517. Epub 2016 May 25. PMID 27216848